CLINICAL TRIAL: NCT03782376
Title: A Phase 3b, Randomized, Double-blind, Multicenter Study to Evaluate the Safety and Efficacy of Intravenous Re-induction Therapy With Ustekinumab in Patients With Moderately to Severely Active Crohn's Disease
Brief Title: A Study to Evaluate Efficacy and Safety of Ustekinumab Re-induction Therapy in Participants With Moderately to Severely Active Crohn's Disease
Acronym: POWER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR108533; 2018-002629-51 (EudraCT Number); CNTO1275CRD3008 (Other: Janssen-Cilag Ltd.)
Record Dates: First submitted 2018-12-11; First posted 2018-12-20 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Ustekinumab (IV re-induction) (Experimental): Participants who experience a secondary loss of response (LoR) to 90 mg ustekinumab maintenance treatment, administered subcutaneously every 8 weeks (q8w) will receive a weight-tiered based ustekinumab IV re-induction dose of approximately 6 mg/kg and matching placebo subcutaneously at Week 0. At Weeks 8 and 16, all participants will receive SC maintenance injections of 90 mg ustekinumab. Participants will resume their standard-of-care therapy at Week 24 at the discretion of the treating physician.
  Interventions: Drug: Ustekinumab approximately 6 mg/kg (IV); Drug: Placebo (SC); Drug: Ustekinumab 90 mg (SC) Group 1
- Group 2: Ustekinumab (Continuous q8w SC maintenance) (Active Comparator): Participants who experience a secondary LoR to 90 mg ustekinumab maintenance treatment, administered subcutaneously q8w will receive ustekinumab 90 mg subcutaneously and matching placebo intravenously at Week 0. At Weeks 8 and 16, all participants will receive SC maintenance injections of 90 mg ustekinumab. Participants will resume their standard-of-care therapy at Week 24 at the discretion of the treating physician.
  Interventions: Drug: Placebo (IV); Drug: Ustekinumab 90 mg (SC) Group 2

INTERVENTIONS:
Drug: Ustekinumab approximately 6 mg/kg (IV) — Participants will receive ustekinumab approximately 6mg/kg intravenously at Week 0.
  Other Names: STELARA
  Arms: Group 1: Ustekinumab (IV re-induction)
Drug: Placebo (SC) — Participants will receive SC injection of placebo at Week 0.
  Arms: Group 1: Ustekinumab (IV re-induction)
Drug: Placebo (IV) — Participants will receive IV infusion of placebo at Week 0.
  Arms: Group 2: Ustekinumab (Continuous q8w SC maintenance)
Drug: Ustekinumab 90 mg (SC) Group 1 — Participants will receive SC injection of ustekinumab 90 mg at Weeks 8 and 16.
  Other Names: STELARA
  Arms: Group 1: Ustekinumab (IV re-induction)
Drug: Ustekinumab 90 mg (SC) Group 2 — Participants will receive SC injection of ustekinumab 90 mg at Weeks 0, 8 and 16.
  Other Names: STELARA
  Arms: Group 2: Ustekinumab (Continuous q8w SC maintenance)

SUMMARY:
The primary purpose of this study is to evaluate the efficacy and safety of a single intravenous (IV) re-induction dose of approximately 6 milligram per kilogram (mg/kg) ustekinumab in participants with secondary loss of response (LoR) to subcutaneous (SC) every 8 Weeks (q8w) 90 mg ustekinumab maintenance therapy.

DETAILED DESCRIPTION:
This study compares the efficacy and safety of a single weight-tiered based IV re-induction dose of approximately 6 mg/kg ustekinumab versus continuing with regular SC q8w 90 mg ustekinumab administration. It consists of screening (5 weeks); treatment period (Week 0 to 24); and safety follow up visit (20 weeks after last dose). The primary hypothesis is that a single IV re-induction dose of ustekinumab is superior to continuing with regular SC q8w maintenance treatment as measured by clinical response after 16 weeks of treatment. Study assessments will include Crohn's disease activity index (CDAI), video ileocolonoscopy, patient-reported outcomes (PROs), laboratory evaluations, biomarkers, review of concomitant medications and adverse events (AEs), and evaluation of serum concentrations of study agent as well as development of antibodies to study agent. All participants will be randomly assigned to receive either ustekinumab IV re-induction or regular SC q8w 90 mg ustekinumab injection at baseline in a double dummy design. No participants will be treated with placebo only.

ELIGIBILITY:
Inclusion criteria:

* A history of Crohn's disease or fistulizing Crohn's disease of at least 3 months' duration, with colitis, ileitis, or ileocolitis, confirmed at any time in the past by radiography, histology, and/or endoscopy
* Currently receiving subcutaneous 90 mg every 8 weeks (q8w) ustekinumab maintenance therapy and initially responded to ustekinumab induction therapy, administered according to the local label, followed by secondary loss of response (LoR) to ustekinumab. Secondary LoR to ustekinumab is defined as active disease at study baseline, proven by a Crohn's Disease Activity Index (CDAI) score of greater than or equal to (>=) 220 and <=450 with at least one of the following: Elevated C-reactive protein (CRP) (>3.0 milligram per liter [mg/L]); and/or elevated Fecal calprotectin (fCal) >250 milligram per kilogram [mg/kg]); and/or endoscopy (performed less than or equal to (<=) 3 months before baseline) with evidence of active Crohn's disease, (defined as one or more ulcerations in the ileum and/or colon)
* Participants receiving either oral 5-aminosalicylic acid (5-ASA) compounds, oral corticosteroids (for example {e.g.}, prednisone, budesonide) at a prednisone-equivalent dose of <=40 mg/day or <=9 mg/day of budesonide, antibiotics used as the primary treatment of Crohn's disease, or conventional immunomodulators (i.e., azathioprine [AZA], 6-mercaptopurine [6-MP], or methotrexate [MTX]) are permitted providing the doses indicated are stable before baseline or have been discontinued before baseline within the protocol defined durations

Exclusion Criteria:

* Complications of Crohn's disease, such as symptomatic strictures or stenoses, short gut syndrome, or any other manifestation that might be anticipated to require surgery, could preclude the use of the CDAI to assess response to therapy, or would possibly confound the ability to assess the effect of treatment with ustekinumab
* Currently has or is suspected to have an abscess. Recent cutaneous and perianal abscesses are not exclusionary if drained and adequately treated at least 3 weeks before baseline (or 8 weeks before baseline for intra-abdominal abscesses) provided there is no anticipated need for any further surgery. Participants with active fistulas may be included if there is no anticipation of a need for surgery and there are currently no abscesses identified
* Any kind of bowel resection within 6 months or any other intra-abdominal surgery within 3 months before baseline
* A draining (i.e., functioning) stoma or ostomy
* Received ustekinumab intravenous re-induction after the initial weight-tiered-based IV induction dose of ustekinumab
* Any known history of shortened frequency of SC dose administration (<q8w) for a secondary loss of response where the participant did not, in the opinion of the treating physician, benefit from the dose interval shortening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2023-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd. Clinical Trial, Study Director — Janssen-Cilag Ltd.
Locations (104):
- United States (28):
  - University of California, San Diego, La Jolla, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Florida Research Network, LLC, Gainesville, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Advent Health, Orlando, Florida
  - Florida Hospital Tampa, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Atlanta Gastroenterology Associates, (AGA) LLC - Emory Saint Joseph's, Atlanta, Georgia
  - Atlanta Gastroenterology Specialists, Suwanee, Georgia
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Brigham And Women's Hospital, Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University School Of Medicine, St Louis, Missouri
  - Mount Sinai School of Medicine, New York, New York
  - Ohio State University Hospital, Hilliard, Ohio
  - Northshore Gastroenterology Research, LLC, Westlake, Ohio
  - Oklahoma Digestive Disease Specialists, Oklahoma City, Oklahoma
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Digestive Disease Consultants, Cedar Park, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Gastroenterology Research of America, LLC, San Antonio, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Washington, Seattle, Washington
  - Washington Gastroenterology, PLLC, Tacoma, Washington
- Austria (2):
  - Krankenhaus der Barmherzigen Brüder, Vienna
  - Medizinische Universitaet Wien, Vienna
- Czechia (2):
  - Hepato-gastroenterologie HK, s.r.o., Hradec Králové
  - ISCARE a.s., Prague
- France (7):
  - Hopital Beaujon, Clichy
  - CHRU de Lille Hopital Claude Huriez, Lille
  - CHRU Montpellier - Hopital Saint-Eloi, Montpellier
  - CHU Hopital Saint Antoine, Paris
  - Hospices Civils de Lyon HCL, Pierre-Bénite
  - CHRU Hopital de Pontchaillou, Rennes
  - CHU de Nancy_ Hopital Brabois, Vandœuvre-lès-Nancy
- Germany (21):
  - Klinikum Augsburg, Augsburg
  - GASTRO-Studien, Berlin
  - Charite - Universitaetsmedizin Berlin (CCM), Berlin
  - Medizinisches Versorgungszentrum (MVZ) Dachau, Dachau
  - University Hospital Dresden, Dresden
  - Agaplesion Frankfurter Diakonie Kliniken GmbH, Markus Krankenhaus, Frankfurt
  - Universitatsklinikum Frankfurt/ Medizinische Klinik 1, Frankfurt
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - Städtisches Krankenhaus Martha-Maria Halle-Dölau gGmbH, Halle
  - Hamburgisches Forschungsinstitut fuer CED, HaFCED e.K., Hamburg
  - Gastroenterologie Opernstrasse, Kassel
  - Universitatsklinikum Schleswig Holstein Kiel, Kiel
  - Staedtisches Klinikum Lueneburg, Lüneburg
  - Universitätsklinikum Otto-von-Guericke-Universität Magdeburg, Magdeburg
  - Medizinische Fakultät Mannheim der Universität Heidelberg, Mannheim
  - Gastroenterologische Gemeinschaftspraxis Minden, Minden
  - Klinikum der Universitaet Muenchen, München
  - Praxis Dr. med. Ulf Helwig, Oldenburg
  - Zentrum für Gastroenterologie Saar MVZ GmbH, Saarbrücken
  - Universitaetsklinik Tuebingen, Tübingen
  - Universitaetsklinikum Ulm, Klinik fuer Innere Medizin II, Ulm
- Italy (6):
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale Villa Sofia-Cervello, Palermo
  - Azienda Ospedaliera G.Salvini Ospedale di Rho, Rho
  - Fondazione Policlinico Gemelli Università Cattolica, Roma
  - Istituto Clinico Humanitas, Rozzano
  - AO Ordine Mauriziano, Torino
- Netherlands (6):
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Leiden University Medical Center, Leiden
  - Maastricht Universitair Medisch Centrum, Maastricht
  - Radboudumc, Nijmegen
  - Erasmus MC, Rotterdam
  - Sint Franciscus Gasthuis, Rotterdam
- Russia (4):
  - Irkutsk State Medical Academy of Postgraduate Education, Irkutsk
  - Olla-Med, Llc, Moscow
  - City Clinical Hospital #31, Saint Petersburg
  - GBUZ Respublican Clinical Hospital n.a. GG Kuvatova, Ufa
- South Korea (5):
  - Inje University Haeundae Paik Hospital, Busan
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - KyungHee University Hospital, Seoul
- Spain (15):
  - Hosp. Univ. Fundacion Alcorcon, Alcorcón
  - Hosp. Arquitecto Marcide, Ferrol
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Hosp Virgen de La Victoria, Málaga
  - Hosp. Univ. Virgen de La Arrixaca, Murcia
  - Hosp. de Navarra, Pamplona
  - Hosp. Montecelo, Pontevedra
  - Corporacio Sanitari Parc Tauli, Sabadell
  - Hosp Clinico Univ de Salamanca, Salamanca
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Hosp. Clinico Univ. de Valencia, Valencia
  - Hosp. Alvaro Cunqueiro, Vigo
  - Hosp. Clinico Univ. Lozano Blesa, Zaragoza
  - Hosp. Univ. Miguel Servet, Zaragoza
- Sweden (2):
  - Gastromottagningen, Malmo
  - Gastromottagningen, Stockholm
- United Kingdom (6):
  - Pennine Acute Hospitals-Fairfield General Hospital, Bury
  - Gloucestershire Hospitals NHS Foundation Trust - Cheltenham, Cheltenham
  - Royal Devon & Exeter Hospital, Exeter
  - King's College Hospital NHS Foundation Trust, London
  - St George's Hospital, London
  - Southampton University Hospitals NHS Trust, Southampton

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials\transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale open and Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Hasskamp J, Meinhardt C, Timmer A. Anti-IL-12/23p40 antibodies for induction of remission in Crohn's disease. Cochrane Database Syst Rev. 2025 May 13;5(5):CD007572. doi: 10.1002/14651858.CD007572.pub4. PMID 40357993
- [Derived] Ten Bokkel Huinink S, Biemans V, Duijvestein M, Pierik M, Hoentjen F, West RL, van der Woude CJ, de Vries AC. Re-induction with intravenous Ustekinumab after secondary loss of response is a valid optimization strategy in Crohn's disease. Eur J Gastroenterol Hepatol. 2021 Dec 1;33(1S Suppl 1):e783-e788. doi: 10.1097/MEG.0000000000002256. PMID 34334713

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Ustekinumab (IV Re-induction): Participants who initially responded to ustekinumab induction therapy followed by a secondary loss of response (LoR) to ustekinumab administered as subcutaneous (SC) injection every 8 weeks (q8w) maintenance therapy received a weight-tiered based re-induction dose of ustekinumab 6 milligrams per kilogram (mg/kg) as an intravenous (IV) infusion and placebo matching to ustekinumab as SC injection at Week 0. At Weeks 8 and 16, all participants received ustekinumab 90 mg maintenance dose as SC injection. At Week 24, all participants underwent study assessments before resuming their standard-of-care therapy at the discretion of the treating physician. Participants were followed-up for safety up to Week 36.
- Group 2: Ustekinumab (Continuous q8w SC Maintenance): Participants who initially responded to ustekinumab induction therapy followed by a secondary LoR to ustekinumab administered as SC injection q8w maintenance therapy received ustekinumab 90 mg as SC injection and placebo matching to ustekinumab as an IV infusion at Week 0. At Weeks 8 and 16, all participants received ustekinumab 90 mg maintenance dose as SC injection. At Week 24, all participants underwent study assessments before resuming their standard-of-care therapy at the discretion of the treating physician. Participants were followed-up for safety up to Week 36.
Period: Overall Study
Arm/Group | Group 1: Ustekinumab (IV Re-induction) | Group 2: Ustekinumab (Continuous q8w SC Maintenance)
Started | 108 | 107
Completed | 82 | 77
Not Completed | 26 | 30
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 7 | 11
Not completed — Death | 1 | 0
Not completed — Other | 16 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Ustekinumab (IV Re-induction) | Group 2: Ustekinumab (Continuous q8w SC Maintenance) | Total
Number analyzed (Participants) | 108 | 107 | 215
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (13.63) | 40 (13.07) | 40.9 (13.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 62 | 124
  Male | 46 | 45 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 103 | 103 | 206
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 10 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 90 | 89 | 179
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 6 | 3 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  Czech Republic | 1 | 4 | 5
  France | 9 | 5 | 14
  Germany | 36 | 33 | 69
  Italy | 6 | 4 | 10
  Netherlands | 1 | 4 | 5
  Republic of Korea | 4 | 7 | 11
  Russia | 3 | 5 | 8
  Spain | 10 | 6 | 16
  Sweden | 1 | 1 | 2
  United Kingdom | 4 | 4 | 8
  United States of America | 33 | 34 | 67

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Response at Week 16
Description: Clinical response was defined as greater than or equal to (>=) 100-point reduction from baseline in Crohn's disease activity index (CDAI) score or a CDAI score < 150 points. CDAI is validated multi-item measure of severity of illness derived as weighted sum of 8 different Crohn's disease (CD)-related variables (extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid stools, abdominal pain/cramping, use of antidiarrheal drug(s) and/or opiates, and general well-being). The last 4 variables were scored over 7 days by participant on diary card. In general, CDAI score ranges from 0 to approximately 600; higher score=higher disease activities. Participants who had prohibited CD-related surgery, prohibited concomitant medication changes or discontinued study agent due to lack of efficacy or adverse event indicated to be of worsening CD prior to designated analysis timepoint were considered not to be in clinical response, regardless of their CDAI score.
Time Frame: Week 16
Population: Full analysis set included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Ustekinumab (IV Re-induction) | Group 2: Ustekinumab (Continuous q8w SC Maintenance)
Number analyzed (Participants) | 108 | 107
Percentage of participants | 49.1 | 37.4
Statistical Analysis 1: Comparison: Group 1: Ustekinumab (IV Re-induction) vs Group 2: Ustekinumab (Continuous q8w SC Maintenance); The fixed sequence testing method was used. CMH chi-square test (2-sided) stratified by baseline CDAI score (<= 300 or > 300), and prior biologic failure status at baseline (yes or no); Test type: Superiority; p = 0.089, Cochran-Mantel Haenszel-chi-square test — Threshold for significance was 0.05 level; Difference in percentage = 11.5, 95% CI 2-sided [-1.5 to 24.5]

2. Secondary Outcome: Percentage of Participants With Clinical Remission at Week 16
Description: Percentage of participants with clinical remission at Week 16 were reported. Clinical remission was defined as CDAI score of <150 points. CDAI is a validated multi-item measure of severity of illness derived as weighted sum of 8 different CD-related variables (extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid stools, abdominal pain/cramping, use of antidiarrheal drug(s) and/or opiates and general well-being). The last 4 variables were scored over 7 days by participant on diary card. In general, CDAI score ranges from 0 to approximately 600; higher score=higher disease activities. Participants who had prohibited CD-related surgery, prohibited concomitant medication changes or discontinued study agent due to lack of efficacy or adverse event indicated to be of worsening CD prior to designated analysis timepoint were considered not to be in clinical remission, regardless of their CDAI score.
Time Frame: Week 16
Population: Full analysis set included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Ustekinumab (IV Re-induction) | Group 2: Ustekinumab (Continuous q8w SC Maintenance)
Number analyzed (Participants) | 108 | 107
Percentage of participants | 33.3 | 27.1
Statistical Analysis 1: Comparison: Group 1: Ustekinumab (IV Re-induction) vs Group 2: Ustekinumab (Continuous q8w SC Maintenance); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.338, CMH chi-square test (2-sided); Difference in percentage = 5.9, 95% CI 2-sided [-6.0 to 17.8]

3. Secondary Outcome: Percentage of Participants With Clinical Response at Week 8
Description: Clinical response was defined as a >=100-point reduction from the baseline in CDAI score or a CDAI score <150 point. The CDAI is a validated multi-item measure of severity of illness derived as a weighted sum of 8 different CD-related variables (extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid stools, abdominal pain/cramping, use of antidiarrheal drug(s) and/or opiates, and general well-being). The last 4 variables were scored over 7 days by the participant on a diary card. In general, CDAI score ranges from 0 to approximately 600; higher score indicates higher disease activities. Participants who had prohibited CD-related surgery, prohibited concomitant medication changes or discontinued study agent due to lack of efficacy or adverse event indicated to be of worsening CD prior to designated analysis timepoint were considered not to be in clinical response, regardless of their CDAI score.
Time Frame: Week 8
Population: Full analysis set included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Ustekinumab (IV Re-induction) | Group 2: Ustekinumab (Continuous q8w SC Maintenance)
Number analyzed (Participants) | 108 | 107
Percentage of participants | 51.9 | 44.9
Statistical Analysis 1: Comparison: Group 1: Ustekinumab (IV Re-induction) vs Group 2: Ustekinumab (Continuous q8w SC Maintenance); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.300, CMH chi-square test (2-sided); Difference in percentage = 7.1, 95% CI 2-sided [-6.0 to 20.2]

4. Secondary Outcome: Percentage of Participants With Clinical Remission at Week 8
Description: Percentage of participants with clinical remission at Week 8 were reported. Clinical remission was defined as CDAI score of <150 points. CDAI is a validated multi-item measure of severity of illness derived as weighted sum of 8 different CD-related variables (extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid stools, abdominal pain/cramping, use of antidiarrheal drug(s) and/or opiates and general well-being). The last 4 variables were scored over 7 days by participant on diary card. In general, CDAI score ranges from 0 to approximately 600; higher score=higher disease activities. Participants who had prohibited CD-related surgery, prohibited concomitant medication changes or discontinued study agent due to lack of efficacy or adverse event indicated to be of worsening CD prior to designated analysis timepoint were considered not to be in clinical remission, regardless of their CDAI score.
Time Frame: Week 8
Population: Full analysis set included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Ustekinumab (IV Re-induction) | Group 2: Ustekinumab (Continuous q8w SC Maintenance)
Number analyzed (Participants) | 108 | 107
Percentage of participants | 35.2 | 29.0
Statistical Analysis 1: Comparison: Group 1: Ustekinumab (IV Re-induction) vs Group 2: Ustekinumab (Continuous q8w SC Maintenance); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.314, CMH chi-square test (2-sided); Difference in percentage = 6.4, 95% CI 2-sided [-5.8 to 18.6]

5. Secondary Outcome: Percentage of Participants With Normalization of C-reactive Protein (CRP) and/or Normalization of Fecal Calprotectin (fCal) Concentration at Week 16
Description: Percentage of participants with normalization at Week 16, among participants with elevated CRP and/or fCal at baseline were reported. Participants were considered to be normalized if at least one biomarker (fCal or CRP) was normalized. Normalized CRP=CRP value less than or equal to (<=) 3 milligrams per liter(mg/L). Normalized fCal concentrations was defined as <=250 micrograms per gram(mcg/g). When either CRP or FCal value was abnormal at baseline and value of same parameter normalizes at designated analysis timepoint, participants were considered to be normalized at designated analysis timepoint. Participants who had prohibited CD-related surgery, prohibited concomitant medication changes, or discontinued study agent due to lack of efficacy or adverse event indicated to be of worsening CD prior to designated analysis timepoint are considered not to be normalized. Participants who had insufficient data at designated analysis timepoint had their last value carried forward.
Time Frame: Week 16
Population: Full analysis set included all randomized participants with either elevated CRP and/or elevated fCal at baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Ustekinumab (IV Re-induction) | Group 2: Ustekinumab (Continuous q8w SC Maintenance)
Number analyzed (Participants) | 93 | 94
Percentage of participants | 33.3 | 14.9
Statistical Analysis 1: Comparison: Group 1: Ustekinumab (IV Re-induction) vs Group 2: Ustekinumab (Continuous q8w SC Maintenance); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.004, CMH chi-square test (2-sided); Difference in percentage = 18.5, 95% CI 2-sided [6.8 to 30.2]

6. Secondary Outcome: Percentage of Participants With Clinical Remission at Week 24
Description: Percentage of participants with clinical remission at Week 24 were reported. Clinical remission was defined as CDAI score of <150 points. CDAI is a validated multi-item measure of severity of illness derived as weighted sum of 8 different CD-related variables (extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid stools, abdominal pain/cramping, use of antidiarrheal drug(s) and/or opiates and general well-being). The last 4 variables were scored over 7 days by participant on diary card. In general, CDAI score ranges from 0 to approximately 600; higher score=higher disease activities. Participants who had prohibited CD-related surgery, prohibited concomitant medication changes or discontinued study agent due to lack of efficacy or adverse event indicated to be of worsening CD prior to designated analysis timepoint were considered not to be in clinical remission, regardless of their CDAI score.
Time Frame: Week 24
Population: Full analysis set included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Ustekinumab (IV Re-induction) | Group 2: Ustekinumab (Continuous q8w SC Maintenance)
Number analyzed (Participants) | 108 | 107
Percentage of participants | 37.0 | 27.1

7. Secondary Outcome: Percentage of Participants With Clinical Response at Week 24
Description: Clinical response was defined as a >=100-point reduction from the baseline in CDAI score or a CDAI score <150 point. The CDAI is a validated multi-item measure of severity of illness derived as a weighted sum of 8 different Crohn's disease-related variables (extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid stools, abdominal pain/cramping, use of antidiarrheal drug(s) and/or opiates, and general well-being). The last 4 variables were scored over 7 days by the participant on a diary card. In general, CDAI score ranges from 0 to approximately 600; higher score indicates higher disease activities. Participants who had prohibited CD-related surgery, prohibited concomitant medication changes or discontinued study agent due to lack of efficacy or adverse event indicated to be of worsening CD prior to designated analysis timepoint were considered not to be in clinical response, regardless of their CDAI score.
Time Frame: Week 24
Population: Full analysis set included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Ustekinumab (IV Re-induction) | Group 2: Ustekinumab (Continuous q8w SC Maintenance)
Number analyzed (Participants) | 108 | 107
Percentage of participants | 47.2 | 39.3

8. Secondary Outcome: Percentage of Participants With Normalization of C-reactive Protein (CRP) and/or Normalization of Fecal Calprotectin (fCal) Concentration at Week 24
Description: Percentage of participants with normalization at Week 24, among participants with elevated CRP and/or fCal at baseline were reported. Participants were considered to be normalized if at least one biomarker (fCal or CRP) was normalized. Normalized CRP=CRP value less than or equal to (<=) 3 milligrams per liter(mg/L). Normalized fCal concentrations was defined as <=250 micrograms per gram(mcg/g). When either CRP or FCal value was abnormal at baseline and value of same parameter normalizes at designated analysis timepoint, participants were considered to be normalized at designated analysis timepoint. Participants who had prohibited CD-related surgery, prohibited concomitant medication changes, or discontinued study agent due to lack of efficacy or adverse event indicated to be of worsening CD prior to designated analysis timepoint are considered not to be normalized. Participants who had insufficient data at designated analysis timepoint had their last value carried forward.
Time Frame: Week 24
Population: Full analysis set included all randomized participants with either elevated CRP and/or elevated fCal at baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Ustekinumab (IV Re-induction) | Group 2: Ustekinumab (Continuous q8w SC Maintenance)
Number analyzed (Participants) | 93 | 94
Percentage of participants | 26.9 | 21.3

9. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An adverse event does not necessarily have a causal relationship with the treatment. TEAEs were adverse events with onset during the intervention phase or that were a consequence of a pre-existing condition that had worsened since baseline. Any AE occurring at or after the initial administration of study agent through the end of the trial was considered to be treatment emergent. In this outcome measure, TEAEs including all AEs irrespective of being serious or non-serious AE are reported.
Time Frame: From baseline (Week 0) up to Week 36
Population: Safety analysis set included all randomized participants who received at least 1 administration of study agent. Participants were analyzed according to the actual treatment received.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Ustekinumab (IV Re-induction) | Group 2: Ustekinumab (Continuous q8w SC Maintenance)
Number analyzed (Participants) | 108 | 107
Percentage of participants | 70.4 | 72.9

10. Secondary Outcome: Percentage of Participants With Treatment-emergent Serious Adverse Events (TESAEs)
Description: A serious adverse event (SAE) was an adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; a suspected transmission of any infectious agent via a medicinal product; medically important. TESAEs were adverse events with onset during the intervention phase or that are a consequence of a pre-existing condition that had worsened since baseline. Any AE occurring at or after the initial administration of study agent through the end of the trial was considered to be treatment emergent.
Time Frame: From baseline (Week 0) up to Week 36
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Ustekinumab (IV Re-induction) | Group 2: Ustekinumab (Continuous q8w SC Maintenance)
Number analyzed (Participants) | 108 | 107
Percentage of participants | 8.3 | 12.1

11. Secondary Outcome: Percentage of Participants With Treatment-emergent Infections
Description: Percentage of participants with treatment-emergent infections were reported. Any infection occurring at or after the initial administration of study agent through the end of the trial was considered to be treatment emergent.
Time Frame: From baseline (Week 0) up to Week 36
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Ustekinumab (IV Re-induction) | Group 2: Ustekinumab (Continuous q8w SC Maintenance)
Number analyzed (Participants) | 108 | 107
Percentage of participants | 33.3 | 29.9

12. Secondary Outcome: Percentage of Participants With Treatment-emergent Serious Infections
Description: Percentage of participants with treatment-emergent serious infections was reported. Any infection occurring at or after the initial administration of study agent through the end of the trial was considered to be treatment emergent.
Time Frame: From baseline (Week 0) up to Week 36
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Ustekinumab (IV Re-induction) | Group 2: Ustekinumab (Continuous q8w SC Maintenance)
Number analyzed (Participants) | 108 | 107
Percentage of participants | 1.9 | 1.9

13. Secondary Outcome: Change From Baseline in Clinical Laboratory Values for Hematology (Hemoglobin) and Chemistry (Albumin, Total Protein)
Description: Change from baseline in clinical laboratory values for hematology (hemoglobin) and chemistry (albumin, total protein) was reported.
Time Frame: Baseline, Weeks 8, 16, 24
Population: Safety analysis set included all randomized participants who received at least 1 administration of study agent. Participants were analyzed according to the actual treatment received. Here, 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure and 'n' (number analyzed) signifies participants who were evaluated at specified timepoints for specified parameters.
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Group 1: Ustekinumab (IV Re-induction) | Group 2: Ustekinumab (Continuous q8w SC Maintenance)
Number analyzed (Participants) | 103 | 98
Grams per liter (g/L)
  Week 8: Hematology (Hemoglobin): number analyzed (Participants) | 103 | 92
  Week 8: Hematology (Hemoglobin) | 2.893 (9.5568) | -0.185 (7.8669)
  Week 16: Hematology (Hemoglobin): number analyzed (Participants) | 94 | 85
  Week 16: Hematology (Hemoglobin) | 3.245 (10.4621) | 0.835 (10.4652)
  Week 24: Hematology (Hemoglobin): number analyzed (Participants) | 74 | 75
  Week 24: Hematology (Hemoglobin) | 3.203 (11.2408) | -0.400 (11.2610)
  Week 8: Chemistry (Albumin): number analyzed (Participants) | 102 | 98
  Week 8: Chemistry (Albumin) | 0.765 (2.9456) | 0.286 (2.6671)
  Week 16: Chemistry (Albumin): number analyzed (Participants) | 97 | 92
  Week 16: Chemistry (Albumin) | 0.567 (3.0649) | 0.554 (3.3753)
  Week 24: Chemistry (Albumin): number analyzed (Participants) | 81 | 77
  Week 24: Chemistry (Albumin) | 0.741 (2.9613) | 0.221 (3.1690)
  Week 8: Chemistry (Total protein): number analyzed (Participants) | 102 | 98
  Week 8: Chemistry (Total protein) | 0.588 (4.6806) | 0.265 (4.3803)
  Week 16: Chemistry (Total protein): number analyzed (Participants) | 97 | 92
  Week 16: Chemistry (Total protein) | 0.340 (5.2418) | 0.783 (4.7690)
  Week 24: Chemistry (Total protein): number analyzed (Participants) | 81 | 78
  Week 24: Chemistry (Total protein) | 0.605 (4.4150) | 0.333 (5.4954)

14. Secondary Outcome: Change From Baseline in Clinical Laboratory Values for Hematology (Hematocrit)
Description: Change from baseline in clinical laboratory values for hematology (hematocrit) was reported.
Time Frame: Baseline, Weeks 8, 16, 24
Population: Safety analysis set included all randomized participants who received at least 1 administration of study agent. Participants were analyzed according to the actual treatment received. Here, 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure and 'n' (number analyzed) signifies participants who were evaluated at specified timepoints.
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells
Arm/Group | Group 1: Ustekinumab (IV Re-induction) | Group 2: Ustekinumab (Continuous q8w SC Maintenance)
Number analyzed (Participants) | 101 | 88
Percentage of red blood cells
  Week 8 | 0.009 (0.0313) | -0.001 (0.277)
  Week 16: number analyzed (Participants) | 90 | 83
  Week 16 | 0.010 (0.0306) | 0.001 (0.0356)
  Week 24: number analyzed (Participants) | 74 | 71
  Week 24 | 0.009 (0.0358) | 0.001 (0.0349)

15. Secondary Outcome: Change From Baseline in Clinical Laboratory Values for Hematology (Total White Blood Cell [WBC], Neutrophils, Absolute Lymphocyte, Eosinophils, Platelets)
Description: Change from baseline in clinical laboratory values for hematology (total WBC, neutrophils, absolute lymphocyte, eosinophils, platelets) was reported.
Time Frame: Baseline, Weeks 8, 16, 24
Population: Safety analysis set included all randomized participants who received at least 1 administration of study agent. Participants were analyzed according to the actual treatment received. Here, 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure and 'n' (number analyzed) signifies participants who were evaluated at specified timepoints for specific parameters.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Group 1: Ustekinumab (IV Re-induction) | Group 2: Ustekinumab (Continuous q8w SC Maintenance)
Number analyzed (Participants) | 103 | 92
10^9 cells/L
  Week 8: Total WBC | -0.386 (1.8358) | -0.272 (1.7301)
  Week 16: Total WBC: number analyzed (Participants) | 94 | 85
  Week 16: Total WBC | -0.329 (2.2700) | -0.124 (2.1404)
  Week 24: Total WBC: number analyzed (Participants) | 74 | 75
  Week 24: Total WBC | -0.149 (2.2347) | 0.104 (1.6612)
  Week 8:Neutrophils | -0.235 (1.7610) | -0.241 (1.6154)
  Week 16: Neutrophils: number analyzed (Participants) | 94 | 85
  Week 16: Neutrophils | -0.195 (2.0172) | -0.053 (2.1811)
  Week 24: Neutrophils: number analyzed (Participants) | 74 | 75
  Week 24: Neutrophils | -0.038 (2.2944) | 0.133 (1.4312)
  Week 8: Absolute Lymphocytes | -0.101 (0.4962) | -0.020 (0.3415)
  Week 16: Absolute Lymphocytes: number analyzed (Participants) | 94 | 85
  Week 16: Absolute Lymphocytes | -0.088 (0.5690) | -0.052 (0.3997)
  Week 24: Absolute Lymphocytes: number analyzed (Participants) | 74 | 75
  Week 24: Absolute Lymphocytes | -0.088 (0.6599) | -0.021 (0.3960)
  Week 8: Eosinophils | -0.009 (0.0876) | -0.004 (0.1153)
  Week 16: Eosinophils: number analyzed (Participants) | 94 | 85
  Week 16: Eosinophils | -0.014 (0.1176) | -0.013 (0.1330)
  Week 24: Eosinophils: number analyzed (Participants) | 74 | 75
  Week 24: Eosinophils | -0.001 (0.0912) | -0.008 (0.1136)
  Week 8: Platelets | -13.65 (56.553) | -0.67 (51.591)
  Week 16: Platelets: number analyzed (Participants) | 93 | 85
  Week 16: Platelets | -13.28 (60.105) | 4.53 (60.785)
  Week 24: Platelets: number analyzed (Participants) | 73 | 73
  Week 24: Platelets | -10.89 (62.671) | -0.53 (56.624)

16. Secondary Outcome: Change From Baseline in Clinical Laboratory Values for Chemistry (Alkaline Phosphatase, Alanine Transaminase [ALT], Aspartate Transaminase [AST])
Description: Change from baseline in clinical laboratory values for chemistry (alkaline, ALT, AST) was reported.
Time Frame: Baseline, Weeks 8, 16, 24
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Units per Liter (U/L)
Arm/Group | Group 1: Ustekinumab (IV Re-induction) | Group 2: Ustekinumab (Continuous q8w SC Maintenance)
Number analyzed (Participants) | 102 | 98
Units per Liter (U/L)
  Week 8: Alkaline Phosphatase | -1.343 (10.7404) | -0.582 (10.3565)
  Week 16: Alkaline Phosphatase: number analyzed (Participants) | 97 | 91
  Week 16: Alkaline Phosphatase | -0.072 (12.9488) | 0.923 (11.5154)
  Week 24: Alkaline Phosphatase: number analyzed (Participants) | 81 | 77
  Week 24: Alkaline Phosphatase | -0.296 (14.2649) | 0.078 (16.1594)
  Week 8: ALT: number analyzed (Participants) | 101 | 97
  Week 8: ALT | -0.347 (9.3642) | -0.412 (7.9001)
  Week 16: ALT: number analyzed (Participants) | 95 | 89
  Week 16: ALT | -0.811 (8.3898) | -0.101 (9.9750)
  Week 24: ALT: number analyzed (Participants) | 80 | 76
  Week 24: ALT | 0.463 (10.1470) | 2.224 (15.5979)
  Week 8: AST: number analyzed (Participants) | 101 | 97
  Week 8: AST | -0.525 (12.0147) | 0.144 (4.8584)
  Week 16: AST: number analyzed (Participants) | 96 | 92
  Week 16: AST | -0.208 (12.6366) | 0.163 (5.4557)
  Week 24: AST: number analyzed (Participants) | 81 | 77
  Week 24: AST | 0.741 (5.6718) | 1.519 (7.3047)

17. Secondary Outcome: Change From Baseline in Clinical Laboratory Values for Chemistry (Total Bilirubin, Direct Bilirubin, Creatinine)
Description: Change from baseline in clinical laboratory values for chemistry (total bilirubin, direct bilirubin, creatinine) was reported.
Time Frame: Baseline, Weeks 8, 16, 24
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: micromole per liter (mcmol/L)
Arm/Group | Group 1: Ustekinumab (IV Re-induction) | Group 2: Ustekinumab (Continuous q8w SC Maintenance)
Number analyzed (Participants) | 102 | 98
micromole per liter (mcmol/L)
  Week 8: Total Bilirubin: number analyzed (Participants) | 101 | 97
  Week 8: Total Bilirubin | 0.639 (2.5303) | -0.131 (2.9617)
  Week 16: Total Bilirubin: number analyzed (Participants) | 97 | 92
  Week 16: Total Bilirubin | 1.476 (3.4135) | 0.555 (3.6679)
  Week 24: Total Bilirubin: number analyzed (Participants) | 81 | 77
  Week 24: Total Bilirubin | 0.687 (3.0396) | 0.254 (3.1664)
  Week 8: Direct Bilirubin: number analyzed (Participants) | 100 | 97
  Week 8: Direct Bilirubin | 0.086 (0.5495) | -0.010 (0.5998)
  Week 16: Direct Bilirubin: number analyzed (Participants) | 92 | 90
  Week 16: Direct Bilirubin | 0.154 (0.6910) | 0.071 (0.7628)
  Week 24: Direct Bilirubin: number analyzed (Participants) | 80 | 76
  Week 24: Direct Bilirubin | 0.109 (0.5393) | 0.009 (0.7612)
  Week 8: Creatinine | -0.446 (8.9118) | -0.308 (9.6489)
  Week 16: Creatinine: number analyzed (Participants) | 97 | 92
  Week 16: Creatinine | 0.624 (9.7987) | 1.117 (9.0316)
  Week 24: Creatinine: number analyzed (Participants) | 81 | 77
  Week 24: Creatinine | 1.717 (9.5267) | 0.336 (8.4020)

18. Secondary Outcome: Change From Baseline in Clinical Laboratory Values for Chemistry (Sodium, Potassium, Chloride, Blood Urea Nitrogen [BUN]/Urea, Calcium, Phosphate)
Description: Change from baseline in clinical laboratory values for chemistry (sodium, potassium, chloride, BUN/urea, calcium, phosphate) was reported.
Time Frame: Baseline, Weeks 8, 16, 24
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Group 1: Ustekinumab (IV Re-induction) | Group 2: Ustekinumab (Continuous q8w SC Maintenance)
Number analyzed (Participants) | 102 | 98
millimoles per liter (mmol/L)
  Sodium: Week 8 | 0.108 (2.5714) | -0.061 (2.2375)
  Sodium: Week 16: number analyzed (Participants) | 97 | 92
  Sodium: Week 16 | -0.165 (2.2299) | 0.011 (2.3370)
  Sodium: Week 24: number analyzed (Participants) | 81 | 77
  Sodium: Week 24 | 0.235 (2.2928) | -0.117 (2.0454)
  Potassium: Week 8: number analyzed (Participants) | 101 | 98
  Potassium: Week 8 | 0.126 (0.3596) | 0.050 (0.3269)
  Potassium: Week 16: number analyzed (Participants) | 97 | 92
  Potassium: Week 16 | 0.105 (0.3745) | -0.002 (0.3933)
  Potassium: Week 24: number analyzed (Participants) | 81 | 77
  Potassium: Week 24 | 0.067 (0.3732) | 0.001 (0.3185)
  Chloride: Week 8 | 0.078 (2.9136) | -0.520 (2.4714)
  Chloride: Week 16: number analyzed (Participants) | 97 | 92
  Chloride: Week 16 | -0.299 (2.4798) | -0.489 (2.5398)
  Chloride: Week 24: number analyzed (Participants) | 81 | 77
  Chloride: Week 24 | 0.160 (2.4107) | -0.481 (2.2160)
  BUN/urea: Week 8 | 0.279 (1.0050) | 0.248 (1.0710)
  BUN/urea: Week 16: number analyzed (Participants) | 97 | 92
  BUN/urea: Week 16 | 0.204 (1.2812) | 0.029 (1.2841)
  BUN/urea: Week 24: number analyzed (Participants) | 81 | 77
  BUN/urea: Week 24 | 0.304 (1.2031) | 0.179 (1.0629)
  Calcium: Week 8 | 0.022 (0.0967) | 0.013 (0.0968)
  Calcium: Week 16: number analyzed (Participants) | 97 | 92
  Calcium: Week 16 | 0.007 (0.1010) | 0.007 (0.1098)
  Calcium: Week 24: number analyzed (Participants) | 81 | 77
  Calcium: Week 24 | 0.008 (0.1101) | 0.004 (0.1109)
  Phosphate: Week 8 | 0.005 (0.2015) | 0.046 (0.2024)
  Phosphate: Week 16: number analyzed (Participants) | 97 | 92
  Phosphate: Week 16 | 0.006 (0.1946) | 0.026 (0.1905)
  Phosphate: Week 24: number analyzed (Participants) | 81 | 77
  Phosphate: Week 24 | 0.018 (0.1612) | 0.021 (0.1938)

ADVERSE EVENTS:
Time Frame: From baseline (Week 0) up to Week 36
Description: Safety analysis set included all randomized participants who received at least 1 administration of study agent. Participants were analyzed according to the actual treatment received.
Arm/Group | Group 1: Ustekinumab (IV Re-induction) | Group 2: Ustekinumab (Continuous q8w SC Maintenance)
All-Cause Mortality (participants affected / at risk) | 1/108 | 0/107
Serious Adverse Events (participants affected / at risk) | 9/108 | 13/107
Other Adverse Events (participants affected / at risk) | 73/108 | 77/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Ustekinumab (IV Re-induction) (N=108) | Group 2: Ustekinumab (Continuous q8w SC Maintenance) (N=107)
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 3
Crohn's Disease (Gastrointestinal disorders) | 1 | 4
Ileal Stenosis (Gastrointestinal disorders) | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 1
Small Intestinal Stenosis (Gastrointestinal disorders) | 1 | 0
Abdominal Abscess (Infections and infestations) | 0 | 1
Anal Abscess (Infections and infestations) | 1 | 1
Tooth Abscess (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Calculus Urinary (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal Atrophy (Renal and urinary disorders) | 0 | 1
Urethral Stenosis (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Ustekinumab (IV Re-induction) (N=108) | Group 2: Ustekinumab (Continuous q8w SC Maintenance) (N=107)
Anaemia (Blood and lymphatic system disorders) | 3 | 2
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 | 2
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Ear Pain (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Eye Irritation (Eye disorders) | 1 | 0
Photophobia (Eye disorders) | 0 | 1
Uveitis (Eye disorders) | 1 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 2 | 1
Abdominal Distension (Gastrointestinal disorders) | 1 | 0
Abdominal Mass (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 5 | 3
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 2
Abdominal Tenderness (Gastrointestinal disorders) | 1 | 0
Anal Eczema (Gastrointestinal disorders) | 0 | 1
Anal Fissure (Gastrointestinal disorders) | 0 | 4
Anal Fistula (Gastrointestinal disorders) | 1 | 0
Anal Skin Tags (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2
Crohn's Disease (Gastrointestinal disorders) | 23 | 29
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Eosinophilic Oesophagitis (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0
Food Poisoning (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Inflammation (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 0
Large Intestine Polyp (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 4
Proctalgia (Gastrointestinal disorders) | 1 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2
Asthenia (General disorders) | 0 | 1
Chills (General disorders) | 0 | 2
Fatigue (General disorders) | 0 | 3
Influenza Like Illness (General disorders) | 2 | 0
Injection Site Erythema (General disorders) | 1 | 1
Injection Site Mass (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 4
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0
Seasonal Allergy (Immune system disorders) | 1 | 0
Abscess Soft Tissue (Infections and infestations) | 1 | 0
Anal Abscess (Infections and infestations) | 1 | 2
Bronchitis (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 12 | 16
Clostridium Difficile Infection (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 1
Coronavirus Infection (Infections and infestations) | 0 | 1
Enteritis Infectious (Infections and infestations) | 0 | 1
Erythema Migrans (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 4
Gastroenteritis Viral (Infections and infestations) | 0 | 1
Gastrointestinal Infection (Infections and infestations) | 1 | 0
Herpes Zoster (Infections and infestations) | 0 | 1
Infected Fistula (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 4 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 5
Otitis Externa (Infections and infestations) | 0 | 1
Pharyngitis Streptococcal (Infections and infestations) | 1 | 0
Pyelitis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 2 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 0
Ureaplasma Infection (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 3 | 3
Vulvovaginal Candidiasis (Infections and infestations) | 0 | 1
Foot Fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 1
Injection Related Reaction (Injury, poisoning and procedural complications) | 0 | 1
Ligament Rupture (Injury, poisoning and procedural complications) | 1 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 1 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 1
Tendon Rupture (Injury, poisoning and procedural complications) | 1 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 1
Vaccination Complication (Injury, poisoning and procedural complications) | 1 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 1
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 2
Blood Creatinine Increased (Investigations) | 1 | 0
Blood Magnesium Decreased (Investigations) | 0 | 1
C-Reactive Protein Increased (Investigations) | 0 | 2
Gamma-Glutamyltransferase Increased (Investigations) | 1 | 0
Sars-Cov-2 Test Positive (Investigations) | 0 | 1
Vitamin D Decreased (Investigations) | 1 | 1
Weight Increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Iron Deficiency (Metabolism and nutrition disorders) | 1 | 0
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1 | 1
Zinc Deficiency (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1
Greater Trochanteric Pain Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rheumatic Disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pituitary Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carotid Arteriosclerosis (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Dizziness Postural (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 8 | 5
Migraine (Nervous system disorders) | 1 | 0
Ophthalmic Migraine (Nervous system disorders) | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 | 0
Affective Disorder (Psychiatric disorders) | 1 | 0
Conversion Disorder (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 2 | 0
Restlessness (Psychiatric disorders) | 1 | 0
Pelvi-Ureteric Obstruction (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 1
Female Genital Tract Fistula (Reproductive system and breast disorders) | 0 | 1
Heavy Menstrual Bleeding (Reproductive system and breast disorders) | 2 | 0
Pelvic Fluid Collection (Reproductive system and breast disorders) | 0 | 1
Scrotal Dermatitis (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tonsillar Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Dermal Cyst (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema Nodosum (Skin and subcutaneous tissue disorders) | 0 | 3
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Superficial Vein Thrombosis (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Some exploratory endpoints including endoscopic assessments for baseline and Week 16, and clinical data for 24 weeks are not reported in this summary and will be included in the manuscript.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will with hold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT03782376/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-17): https://cdn.clinicaltrials.gov/large-docs/76/NCT03782376/SAP_001.pdf